CLINICAL TRIAL: NCT01767662
Title: Natural History and Effectiveness of Parents' Manipulation in Newborn With Talipes Calcaneovalgus,a Randomized Controlled Trial
Brief Title: Effectiveness of Parents' Manipulation in Newborn With Talipes Calcaneus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: si319/2011
Record Dates: First submitted 2013-01-11; First posted 2013-01-14 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Talipes Calcaneovalgus
Keywords: TCV
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- manipulation (Experimental): home program for parents manipulation
  Interventions: Procedure: manipulation
- observe (Placebo Comparator): observation
  Interventions: Procedure: No intervention

INTERVENTIONS:
Procedure: manipulation — home programme
  Arms: manipulation
Procedure: No intervention — observation
  Arms: observe

SUMMARY:
The purpose of this study is to determine effectiveness of parents' manipulation in newborn with talipes calcaneovalgus over observation group.

DETAILED DESCRIPTION:
Talipes calcaneovalgus is one of the common foot deformity in newborn. Most of patients can be cure without specific treatment. Manipulation was easy method that parents can preform by their own and may be beneficial in speeding resolution of deformity.

ELIGIBILITY:
Inclusion Criteria:

* all newborn with talipes calcaneovalgus

Exclusion Criteria:

* patient associated with congenital musculoskeletal anomaly
* patient with other serious medical condition

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-06 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
percent of success treatment with in six month | six month

SECONDARY OUTCOMES:
duration from start treatment until cure | six month

OTHER OUTCOMES:
failure of treatment | six month

CONTACTS AND LOCATIONS:
Overall Officials: Kamolporn Kaewpornsawan, MD,Ph.D, Principal Investigator — Department of orthopaedic surgery Faculty of medicine siriraj hospital Bangkok Thailand
Locations (1):
- Faculty of Medicine Siriraj Hospital Mahidol University, Bangkok, Bangkok, Thailand